CLINICAL TRIAL: NCT03542344
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 1015550 in Healthy Japanese Male Subjects (Double-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: This Study is Done in Healthy Japanese Volunteers. It Looks at How Different Doses of BI 1015550 Are Taken up in the Body and How Well They Are Tolerated.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1305-0017
Record Dates: First submitted 2018-05-17; First posted 2018-05-31 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — BI 1015550

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BI 1015550 12mg (Experimental)
  Interventions: Drug: BI 1015550 6 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BI 1015550 24mg (Experimental)
  Interventions: Drug: BI 1015550 6 mg

INTERVENTIONS:
Drug: BI 1015550 6 mg — Single rising oral dose
  Other Names: Nerandomilast; JASCAYD®
  Arms: BI 1015550 12mg; BI 1015550 24mg
Drug: Placebo — Single rising oral dose
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of BI 1015550 in healthy male subjects following oral administration of single rising doses.

Secondary objectives are the exploration of the pharmacokinetics (PK) including dose proportionality of BI 1015550 after single dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 20 to 45 years (incl.) at screening.
* Body Mass Index (BMI) of 18.5 to 25.0 kg/m2 (incl.) at screening.
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm) at screening
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance at screening
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders, including but not limited to mood disorders and any history of suicidality
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections including viral hepatitis, human immunodeficiency virus (HIV) and/or syphilis. (Subject with positive Hepatitis B core antibody will not allowed to participate in this trial)
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (consumption of more 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Male subjects who do not agree to minimize the risk of female partners becoming pregnant from the first dosing day until three months after the study completion.

Acceptable methods of contraception comprises barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device or hormonal contraceptive since at least two months)

In addition, the following trial-specific exclusion criteria apply:

* Positive or missing fecal occult blood (no retest allowed) at screening
* Positive testing for fecal calprotectin (retest allowed) at screening
* Positive testing for hematuria if confirmed by microscopic urine analysis (retest allowed) at screening
* Any lifetime history of suicidal behavior (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases(in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized, parallel, placebo-controlled and double-blind trial tested single dose of BI 1015550 in 2 rising dose groups (12 and 24 mg). Subjects stayed in-house for 2 days (d) after single oral dose of trial drug and the end of trial examination took place 7 to 8 d after trial drug administration.
Pre-assignment Details: All subjects were screened for eligibility to participants in the trial. Subjects attended specialist sites which would then ensure that they met all strictly implemented inclusion/exclusion criteria. Subjects were not to be assigned to treatment groups if any one of the specific entry criteria were violated.
Groups:
- Placebo: Comparator product: Matching placebo. The medication was administrated orally with about 240 milliliter (mL) of water after an overnight fast of at least 10 hours. 2 subjects from BI 1015550 12 milligram (mg) arm and 2 subjects from BI 1015550 24mg arm taking Placebo are combined.
- BI 1015550 12mg: 2 film-coated tablets with 6mg of BI 1015550 each (12mg total) were administrated as single oral dose with about 240 mL of water after an overnight fast of at least 10 hours.
- BI 1015550 24mg: 4 film-coated tablets with 6mg of BI 1015550 each (24mg total) were administrated as single oral dose with about 240 mL of water after an overnight fast of at least 10 hours.
Period: Overall Study
Arm/Group | Placebo | BI 1015550 12mg | BI 1015550 24mg
Started | 4 | 6 | 6
Completed | 4 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This subject set included data from all subjects who received at least 1 dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 1015550 12mg | BI 1015550 24mg | Total
Number analyzed (Participants) | 4 | 6 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.5 (4.7) | 32.8 (9.3) | 28.7 (8.3) | 29.9 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 4 | 6 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 6 | 6 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 6 | 6 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Drug-related Adverse Events
Description: Number of participants with drug-related adverse events is presented.
Time Frame: From drug administration until end of study, up to 9 days
Population: Treated set (TS): This subject set included data from all subjects who received at least 1 dose of trial drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BI 1015550 12mg | BI 1015550 24mg
Number analyzed (Participants) | 4 | 6 | 6
Participants | 0 | 0 | 0

2. Secondary Outcome: Area Under the Concentration-time Curve of the BI 1015550 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-inf)
Description: Area under the concentration-time curve of the BI 1015550 in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf) is presented.
Time Frame: Within 3 hours before and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 34, 48, 72, 96, 120 hours after drug administration.
Population: Pharmacokinetic parameter analysis set (PKS): This subject set included data from all subjects from the TS who provided at least 1 secondary pharmacokinetic endpoint (AUC0-inf or Cmax) that was not excluded due to a protocol deviation relevant to the evaluation of pharmacokinetics, or due to pharmacokinetic non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hours per Litre (nmol*h/L)
Arm/Group | BI 1015550 12mg | BI 1015550 24mg
Number analyzed (Participants) | 6 | 6
nanomole*hours per Litre (nmol*h/L) | 2410 (20.8) | 5760 (21.6)

3. Secondary Outcome: Maximum Measured Concentration of the BI 1015550 in Plasma (Cmax)
Description: Maximum measured concentration of the BI 1015550 in plasma (Cmax) is presented.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole per Litre (nmol/L)
Arm/Group | BI 1015550 12mg | BI 1015550 24mg
Number analyzed (Participants) | 6 | 6
nanomole per Litre (nmol/L) | 449 (19.1) | 944 (43.5)

ADVERSE EVENTS:
Time Frame: "All-Cause Mortality", "Serious Adverse Events" and "Other Adverse Events": From first drug administration until end-of-study examination, up to 9 days.
Description: Treated set (TS): This subject set included data from all subjects who received at least 1 dose of trial drug.
Groups:
- BI 1015550 Total: The group consists of 6 participants from BI 1015550 12mg arm and 6 participants from BI 1015550 24mg arm taking trial medication.
Arm/Group | Placebo | BI 1015550 12mg | BI 1015550 24mg | BI 1015550 Total
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 1/4 | 0/6 | 0/6 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4) | BI 1015550 12mg (N=6) | BI 1015550 24mg (N=6) | BI 1015550 Total (N=12)
Occult blood positive (Investigations) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The planned 36mg dose was not investigated and dose proportionality was not assessed as the pharmacokinetic variables (Cmax and AUC0-inf) would be higher than the predetermined safety margin with 36mg dose based on the interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT03542344/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT03542344/SAP_001.pdf